CLINICAL TRIAL: NCT07111936
Title: Evaluating the Impact of CONNECT, a Novel Smoking Cessation Intervention, in a Diverse, Multilingual Population
Brief Title: Evaluating the Impact of CONNECT in a Multilingual Population
Acronym: CONNECT-ML
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 25635; NCI-2025-05153 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation; Smoking Cessation Counseling Ability and Practice; Smoking Cessation Counselling; Lung Cancer Screening
Keywords: Multilingual
MeSH Terms: conditions — Smoking Cessation | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in the focus group. Once completed, new participants will be enrolled in the beta group. After interim analysis has been completed, new participants will be enrolled in the randomized arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Focus Group (Other): Participants in the focus group will be interviewed by the study staff and discuss barriers and facilitators to smoking cessation to be implemented in the beta and randomized phases of the study.
  Interventions: Other: Interview
- Beta Group (Active Comparator): Participants will be testing the CONNECT multilingual smoking cessation materials and provide feedback to investigators. Participation will be limited to about 1.5 - 2 hours.
  Interventions: Behavioral: CONNECT Intervention for multilingual populations
- Group 1: CONNECT Multi-lingual intervention (Experimental): Participants receive the CONNECT multilingual smoking cessation intervention finalized in the beta group analysis, that includes multi-lingual interactive video doctor intervention, text messages once weekly for 12 weeks, and several telephone counseling calls. Participants also receive access to a pharmacist to receive counseling about quitting smoking and may prescribe nicotine replacement therapy. Participants will be asked to provide a saliva sample at the end of the study
  Interventions: Behavioral: CONNECT Intervention for multilingual populations; Other: Saliva Sample
- Group 2: Control Group (Experimental): Participants will receive usual care for smoking cessation at routine medical visit and be asked to complete a total of four brief follow-up phone surveys. Participants will be asked to provide a saliva sample at the end of the study.
  Interventions: Other: Saliva Sample

INTERVENTIONS:
Behavioral: CONNECT Intervention for multilingual populations — The program includes interactive Video Doctor visits to provide participants with information tailored to their individual responses and outreach via brief telephone calls and text messaging to follow-up and connect smokers with evidence-based resources for smoking cessation.
  Other Names: CONNECT Multilingual program
  Arms: Beta Group; Group 1: CONNECT Multi-lingual intervention
Other: Saliva Sample — Undergo saliva collection
  Other Names: Saliva Sample collection
  Arms: Group 1: CONNECT Multi-lingual intervention; Group 2: Control Group
Other: Interview — Attend a focus group
  Arms: Focus Group

SUMMARY:
This study aims to broaden the reach of the lung cancer screening (LCS) CONNECT program (NCT04149249, NCT06213532), by developing a version of the program to be available to multilingual communities. The CONNECT program encourages individuals who are undergoing lung cancer screening to also quit smoking by providing a personalized program which includes a video doctor with personalized responses, text message and telephone call support and connection with a pharmacist to assist in obtaining nicotine replacement medication. This clinical trial will develop and ultimately test how well the CONNECT Multilingual (CONNECT ML) program works to improve smoking cessation among current adult smokers within the Spanish and Cantonese speaking communities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Culturally adapt, translate, improve and fine tune the multi-faceted CONNECT program for multilingual smokers

II. Evaluate the CONNECT multilingual program for current smokers in multilingual communities.

III. Assess the impact of the CONNECT Multilingual program on smoking cessation rates and participant utilization of evidence-based resources to help quit smoking

OUTLINE:

FOCUS GROUP (N=24):

Three focus groups, one each with English, Spanish and Cantonese speaking participants (8 in each group) will be led by investigators. Interviews will be recorded, transcribed and translated. Translation of the Spanish and Cantonese transcripts will be done by University of California, San Francisco (UCSF) translation services.

BETA GROUP (N=15):

The investigators will conduct a pilot, beta testing of the intervention materials with English, Spanish and Cantonese speaking participants. Additional feedback and input from the participants will be used to fine tune the CONNECT smoking cessation intervention to be implemented in a randomized trial.

RANDOMIZED CONTROLLED TRIAL (N=400):

Newly enrolled participants will be assigned to 1 of 2 conditions.

* Group 1: Participants receive the CONNECT Multilingual intervention. Participants will be followed up at 1-week, 1-, 3-, and 6-months after treatment assignment. At 6-months, participants will be asked to complete and return an at-home saliva kit to verify their smoking status.
* Group 2: Participants receive usual care from providers at a regular primary care appointment. Participants will be followed up at 1-week, 1-, 3-, and 6-months after treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years old.
* Current smokers defined at smoking at least one cigarette in past 7 days AND eligible for lung cancer screening (LCS) based on smoking history (>=20 pack year history)
* California (CA) residents
* Able to understand and comply with study procedures for the entire length of the study.
* Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Non-smokers.
* Individuals with a diagnosis of lung cancer.
* Individuals receiving hospice care.
* Individuals whose providers do not think that they should participate (e.g., psychiatric illness or significant cognitive impairment that would impede the individuals ability to participate).
* Hearing and/or vision disabilities that would prevent participants from adequately receiving treatment components such as video or telephone counseling.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 439 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants Smoking cessation rates (Randomized groups only) | Up to 6 months
  The rate of smoking cessation will be defined as the percentage of participants who are abstinent from smoking through self-report and biochemical verification using salivary cotinine levels obtained at 6 months after lung cancer screening
Mean number of quit attempts over time (Randomized groups only) | Up to 6 months
  The number of self-reported 7-day quit attempts over time since lung cancer screening (LCS) will be recorded. Mean and standard deviation will be reported.
Percentage of participants who reported use of smoking cessation resources (Randomized groups only) | Up to 6 months
  Self-reported use of evidence-based smoking cessation resources (enabling factors) after the lung cancer screening (for example, pharmacotherapy for smoking cessation, calling the California Smokers Helpline, group or individual counseling from healthcare providers, etc.) will be reported as a percentage of all participants by arm.

SECONDARY OUTCOMES:
Changes in frequency of response to "Are you seriously thinking of quitting smoking?" over time (Randomized groups only) | Up to 6 months
  The participants readiness to quit will be measured using the Stages of Change questionnaire - single item, which asks "Are you seriously thinking of quitting smoking?" Answers range from 'Yes, within the next 30 days', 'Yes, within the next 6 months', and 'No, not thinking of quitting'. Changes in frequency of response over time will be reported.
Changes in scores on the Readiness and Motivation to Quit Smoking Questionnaire (RMQ) over time (Randomized groups only) | Up to 6 months
  The RMQ is a 11 item self-report, that is used to assess the degree to which measures a person may be ready or motivated to change smoking habits and behaviors. The questionnaire consists of 3 factors: Change smoking behavior (5 items), Motivation to cut down (4 items), and Confidence (2 items). Questions are responded to as Yes/No, or range from "Not at all" to "Very", or ask the duration of time before quitting smoking. The greater the number of positive responses indicates a greater readiness to quit, a greater motivation to quit, and/or a greater confidence to quit smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Walsh, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No